CLINICAL TRIAL: NCT02452346
Title: Phase II Clinical Study of the Clinical Efficacy and Safety of Tosedostat in Atients With Myelodysplastic Syndromes (MDS) After Failure of Hypomethylating Agent-Based Therapy
Brief Title: Study of Clinical Efficacy and Safety of Tosedostat in MDS
Acronym: IST-CTI-MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1409015482
Record Dates: First submitted 2015-01-28; First posted 2015-05-22 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — tosedostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Patients (Experimental): Tosedostat 120 mg PO once daily will be administered.
  Interventions: Drug: Tosedostat

INTERVENTIONS:
Drug: Tosedostat — 120 mg PO once daily continuously for each 28 day treatment cycle
  Other Names: CHR-2797

SUMMARY:
Study WCMC IST-CTI-MDS evaluates the safety and tolerability of tosedostat in adult patients with pathologically confirmed MDS (< 20% blasts in bone marrow, peripheral blood, or both) by World Health Organization (WHO) classification after failure of hypomethylating agent-based therapy.

DETAILED DESCRIPTION:
This is a single-center, open label, two-arm phase II study of clinical activity of tosedostat in adult patients with MDS who have failed prior hypomethylating agent-based therapy. Arm A is defined as Revised International Prognostic Scoring Systems (IPSS-R) very low, low, and intermediate disease. Arm B is defined as IPSS-R high or very high risk disease. The two arms are separate and will enroll simultaneously. The dose of tosedostat will be 120 mg once a day continuously for each 28 day treatment cycle. Patients will be assessed for disease response, on average, every two cycles as defined in the protocol. If patient has no response as defined by the protocol after two cycles, azacitidine 75 mg/m2 SC or IV for 5 days may be combined with tosedostat, at the investigator's discretion.The primary endpoint the study is to evaluate the safety and efficacy of tosedostat in two groups of patients with myelodysplastic syndrome who have relapsed after or are refractory or intolerant to azacitidine or decitabine. The primary endpoint for patients with IPSS-R very low, low and intermediate disease is transfusion independence and the primary endpoint for patients with high or very high risk disease is overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and to provide written informed consent
2. At least 18 years of age with pathologically confirmed MDS (<20% blasts in bone marrow, peripheral blood, or both) within 6 weeks prior to screening by WHO classification
3. Must have received at least 4 cycles of decitabine-based or 6 cycles of azacitidine-based therapy and are either refractory to, relapsed after or intolerant to prior therapy with either agent.

   * Primary failure/refractory: Stable or worsening disease after a minimum of 4 cycles of decitabine-based or 6 cycles of azacitidine-based therapy
   * Secondary failure/relapse: Bone marrow blast count increase or loss of hematologic response after initial treatment response with hypomethylating agent-based therapy
   * Intolerance: Intolerance of hypomethylating agent-based therapy regardless of number of cycles completed and clinical response
4. Progression (according to 2006 IWG criteria) at any time after initiation of subcutaneous or intravenous azacitidine or decitabine treatment per labeling during the past 2 years, defined as follows:

   * For patients with <5% BMBL, ≥ 50% increase in BMBL to >5% BMBL
   * For patients with 5-10% BMBL, ≥ 50% increase in BMBL to >10% BMBL
   * For patients with 10-20% BMBL, ≥ 50% increase in BMBL to >20% BMBL
   * For patients with 20-30% BMBL, ≥ 50% increase in BMBL to >30% BMBL
   * Any of the following:
   * ≥ 50% decrease from maximum remission/response levels in granulocytes or PLT
   * Decrease in Hgb concentration by ≥2 g/dL
   * Transfusion dependence, defined as administration of at least 4 RBC units in the past 8 weeks before Screening (patients must have Hgb values < 9 g/dL prior to transfusion to be considered), in the absence of another explanation.
5. Has failed to respond to, relapsed following, not eligible, or opted not to participate in BM transplantation
6. Patients with very low, low or intermediate risk MDS by the IPSS-R must be transfusion-dependent, with a packed red blood cell requirement of ≥ 2 units/month
7. Off azacitidine or decitabine for at least 2 weeks, off all other treatments for MDS for at least 4 weeks. Filgrastim (G-CSF) and EPO are allowed before and during the study as clinically indicated
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
9. Subjects must have adequate hepatic and renal function including the following:

   * Total bilirubin ≤ 1.5 x upper limit of normal (in the absence of Gilbert's syndrome)
   * AST and ALT ≤ 2.5 x upper limit of normal
   * Serum creatinine ≤ 1.5 x upper limit of normal
10. Must have acceptable recovery from clinically significant non-hematologic toxicity after prior therapy.
11. Must have a life expectancy of at least 2 months
12. Screening left ventricular ejection fraction (LVEF) greater than 50% as documented by transthoracic echocardiogram (TTE)
13. Female subject of child-bearing potential and male subjects with female partners of reproductive potential must use acceptable contraceptive methods (hormonal or barrier method of birth control; abstinence) for the duration of time on study and continue to do so for a further 3 months after the end of tosedostat treatment. Should a female subject become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
14. Able to comply with all study procedures during the study including all visits and tests
15. Willing to adhere to the prohibitions and restrictions specified in this protocol
16. Patient must sign an informed consent form (ICF) indicating that s/he understands the purpose of and procedures required for the study and is willing to participate.

Exclusion Criteria:

1. Presence of AML (≥20% blasts in bone marrow, peripheral blood, or both)
2. Presence of serious illness, medical condition, or other medical history, involving the heart, kidney, liver, or other organ system, including abnormal laboratory parameters, which, in the opinion of the Investigator, would be likely to interfere with a subject's participation in the study or with the interpretation of the results.
3. Have known active central nervous system disease or active, uncontrolled, clinically significant infection(s)
4. Have other active malignancies (including other hematologic malignancies) or other malignancies within 12 months before enrollment, except non-melanoma skin cancer or cervical intraepithelial neoplasia
5. Are receiving any other investigational therapy or protocol-prohibited therapy
6. Have received previous treatment with tosedostat
7. Pregnant or breastfeeding females
8. Any prior or co-existing medical condition that in the Investigator's judgment will substantially increase the risk associated with the subject's participation in the study
9. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures
10. Significant* cardiovascular disease defined as:

    * Active heart disease including myocardial infarction within 6 months prior to study entry
    * Symptomatic coronary artery disease
    * Uncontrolled or clinically significant arrhythmia, angina, congestive heart failure
    * Presence of clinically significant valvular heart disease
    * Presence of clinically significant conduction defect on screening ECG
    * Uncontrolled hypertension (i.e., systolic BP >160mmHg, diastolic >90 mmHg in repeated measurements) despite adequate therapy
    * Clinically significant atrial fibrillation * Grade 3/4 in the CTCAE v4.0 grading would generally be considered clinically significant, although this remains a judgment for the Investigator to make.
11. LVEF ≤ 50%
12. Baseline troponin I and b-type natriuretic peptide > Grade I
13. Prior exposure cardiotoxic agent, such as anthracycline, within 3 months of enrollment
14. Concomitant use of drugs that prolong QT/QTc interval except antibiotics, antifungals, and other antimicrobials used as standard of care for the treatment and prevention of infection and/or other such drugs clinically indicated for patient care. When use of concomitant medications with QT-prolonging potential is necessary, ECG must be repeated 4 hours post-dose on Day 1, on Day 3, and on Day 7, and as clinically indicated, relative to start of agent with QT-prolonging potential.
15. Gastrointestinal disorders that may interfere with absorption of drug
16. Active serious infection or sepsis
17. Clinically significant interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Roboz, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee S, Desai P, Edirisinghe B, Pianello S, Curcio T, Samuel M, Ritchie EK, Roboz GJ. Phase II study of the clinical efficacy and safety of tosedostat in patients with myelodysplastic syndromes (MDS) after failure of hypomethylating agent-based therapy. Leuk Lymphoma. 2021 Feb;62(2):498-500. doi: 10.1080/10428194.2020.1832674. Epub 2020 Oct 10. No abstract available. PMID 33043735

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 12
Completed | 3
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 72 [61 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Over All Survival
Description: Survival following treatment to the date of death, assessed up to a period of 3-4 years.
Time Frame: from start of treatment until death, assessed up to a period of 3-4 years.
Measure: Median (Full Range); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 12
months | 15.9 [2.5 to 30.7]

2. Secondary Outcome: Overall Response
Description: Overall response according to IWG 2006 criteira
Time Frame: Approximately 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 12
Participants
  Complete Remission | 1
  Stable Disease | 8
  Non-evaluable | 3

3. Secondary Outcome: One Year and Two Year Survival
Time Frame: from start of treatment to 1 year and 2 years post treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 12
Participants
  One year survival | 8
  two year survival | 4

ADVERSE EVENTS:
Time Frame: The adverse event data was collected for a period of approx. 3 years from the date of enrollment.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 9/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Other - Decline in performance status (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Fever (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=12)
Other - BNP increased (Investigations) | 7
Electrocardiogram QT corrected interval prolonged (Investigations) | 6
Fatigue (General disorders) | 6
Bruising (Injury, poisoning and procedural complications) | 5
Diarrhea (Gastrointestinal disorders) | 5
Edema limbs (General disorders) | 5
Hypomagnesemia (Investigations) | 4
Alanine transferase increased (Investigations) | 3
Dizziness (Nervous system disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Ejection fraction decreased (Investigations) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Platelet count decreased (Investigations) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
GGT increased (Investigations) | 2
Insomnia (Psychiatric disorders) | 2
Neutrophil count decreased (Investigations) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Alkaline phosphatase increased (Investigations) | 1
Allergic reaction (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Blurred vision (Eye disorders) | 1
Cardiac troponin I increased (Investigations) | 1
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Edema face (General disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
INR increased (Investigations) | 1
Lethargy (Nervous system disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neuralgia (Nervous system disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Other - Demand ischemia (Cardiac disorders) | 1
Other - Ferritin increased (Investigations) | 1
Other - Forgetfulness (Psychiatric disorders) | 1
Other - left subconjunctival hemorrhage (Eye disorders) | 1
Other - Lip excoriation (Injury, poisoning and procedural complications) | 1
Other - Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Other - Muscle spasm (Musculoskeletal and connective tissue disorders) | 1
Other - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Paresthesia, foot (Nervous system disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT02452346/Prot_SAP_000.pdf